CLINICAL TRIAL: NCT03515148
Title: Effectiveness of Eccentric Exercise With a Vibration Program Versus Cryotherapy in Rectus Abdomini Muscle Thickness and Inter-recti Distance in Patients With Chronic Mid Portion Achilles Tendinopathy: A Randomized Clinical Trial
Brief Title: Effectiveness of EE With Vibration Versus Cryotherapy in Rectus Abdomini Muscle Thickness and Inter-recti Distance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Pedro Javier Martin, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tendon02
Record Dates: First submitted 2018-04-21; First posted 2018-05-03 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Achilles Tendinopathy; Diastasis Recti
Keywords: Achilles Tendinopathy; Rectus Abominis; Vibration; Cryotherapy; Eccentric Exercise
MeSH Terms: interventions — Cryotherapy; Vibration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy and eccentric exercise (Experimental): 12 weeks, 5 days/week, once a day, 2 exercise, 3 sets/execise, 15 repetition/set of eccentric exercise of foot plantar flexors First exercise with knee in extension, second exercise with knee in flexion. Previously subjects should cold their leg in ice water during sexteen minutes at a temperature of 8ºC (+/-2ºC)
  Interventions: Procedure: Cryotherapy and eccentric exercise
- Vibration and eccentric exercise (Experimental): 12 weeks, 5 days/week, once a day, 2 exercise, 3 sets/execise, 15 repetition/set of eccentric exercise of foot plantar flexors First exercise with knee in extension, second exercise with knee in flexion.During the exercise subjects will be subjected to vibration. Vibrations parameters: Frequency: 35Hz, Amplitude: 4 milimeters, Force: 3,9G
  Interventions: Procedure: Vibration and eccentric exercise

INTERVENTIONS:
Procedure: Cryotherapy and eccentric exercise — 12 weeks, 5 days/week, once a day, 2 exercise, 3 sets/execise, 15 repetition/set of eccentric exercise of foot plantar flexors First exercise with knee in extension, second exercise with knee in flexion. Previously subjects should cold their leg in ice water during sexteen minutes at a temperature of 8ºC (+/-2ºC)
  Arms: Cryotherapy and eccentric exercise
Procedure: Vibration and eccentric exercise — 12 weeks, 5 days/week, once a day, 2 exercise, 3 sets/execise, 15 repetition/set of eccentric exercise of foot plantar flexors First exercise with knee in extension, second exercise with knee in flexion.During the exercise subjects will be subjected to vibration. Vibrations parameters: Frequency: 35Hz, Amplitude: 4 milimeters, Force: 3,9G
  Arms: Vibration and eccentric exercise

SUMMARY:
The purpose of this study is to determinate de efectiveness of eccentric exercise combined with vibration or cryotherapy in achilles tendinopathy and its effects on the anterior rectus abdominis muscle.

The investigators hypothesis is the combined eccentric exercise with vibration get better results than cryotherapy with eccentric exercise in rectus abdominis muscle parameters.

ELIGIBILITY:
Inclusion Criteria:

* Sports people
* Positive initial ultrasound diagnosis
* Presence of degenerative changes at achilles mid portion
* Chronic Achilles tendon pain, (3/10 VAS)
* Pain when walking or running of Achilles tendon, (3/10 VAS)
* Pain in load in plantar flexion of Achilles tendon, 3/10 VAS)
* Pain in palpation of Achilles, (3/10 VAS)
* Morning Stiffness

Exclusion Criteria:

* Receive physical, orthotic or physiotherapeutic treatment
* Asociated low back pain, ankle/knee/hip injury that may affect the study
* Previous injury or surgery of Achilles tendon.
* Pathologies that may limit the joint of ankle
* Pregnancy
* Obesity
* Patients with diabetes and/or other endocrine or metabolic pathologies or neurologic pathologies
* Patients diagnosed with cardiovascular disease
* Subjets diagnosed with familiar hypercholesterolemia and/or presence of xanthomas or with hyperuricemia
* Patients who have received renal transplantation
* Subjects who have suffered retinal detachment
* Subjects who have received oral contraceptives, statins, corticoids or hormone replacement therapy in the last six months
* Subjects who have received treatment wiht fluoroquinolones in the last two years
* Subjects who have received treatment with AINE's in the last four weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Inter-recti distance | 3 months
  Ultrasound diagnosis
Rectus abdominis thickness | 3 months
  Ultrasound diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Martin, Principal Investigator — Pejamalla@gmail.com
Locations (1):
- Universidad Europea, Madrid, Spain